CLINICAL TRIAL: NCT04844437
Title: Intrapartum Translabial Ultrasonography Reliability in Comparison With Traditional Digital Examination
Brief Title: Intrapartum Translabial Ultrasonography Reliability
Acronym: ITUSR
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sehit Prof. Dr. Ilhan Varank Sancaktepe Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Arzu Bilge Tekin, Specialist, Sehit Prof. Dr. Ilhan Varank Sancaktepe Training and Research Hospital
Other Study IDs: ITUSR
Record Dates: First submitted 2021-04-10; First posted 2021-04-14 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Labour;Obstructed; Progression; Delivery Problem for Fetus; Ultrasound Therapy; Complications
Keywords: labor; intrapartum ultrasonography; head station
MeSH Terms: conditions — Dystocia; Disease Progression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Digital examination of fetal head decent in pregnant women: Pregnant women at 36 weeks or over gestational age in the active phase of the first stage or second stage of labor were examined by digital examination and fetal head station evaluated by two clinicians.
- Transperineal assessment of fetal head decent in pregnant women: Pregnant women at 36 weeks or over gestational age in the active phase of the first stage or second stage of labor were examined by transperineal ultrasound and fetal head station evaluated by two experienced clinicians.
  Interventions: Diagnostic Test: Transperineal ultrasound

INTERVENTIONS:
Diagnostic Test: Transperineal ultrasound — The fetal head station is evaluated by transperineal ultrasonography in valsalva.
  Groups: Transperineal assessment of fetal head decent in pregnant women

SUMMARY:
In a present study vaginal examination of the fetal head station is compared with transperineal ultrasonography evaluation of fetal head station and the ability of ultrasonography evaluation in predicting the time and mode of delivery will be investigated.

DETAILED DESCRIPTION:
The sonographically measured head station, 'ITU station', was measured along the longest visible axis of the fetal head, between the intersections with the infra pubic line and the deepest bony part of the fetal head, subtracting 3 cm for the level of the ischial spines. This parameter is useful to determine the level of engagement of the fetal head and its progression throughout labor.

The labor is divided into a latent phase (stage 0), an active phase (stage 1 and 2), and a third stage defined as the time period between the delivery of the baby and the delivery of the placenta. According to the classic definition, the onset of labor is when regular contractions have been established. The latent phase is characterized by painful contractions and cervical dilatation up to 5 cm in accordance with WHO.

The fetal descent in the birth canal is assessed by vaginal digital examinations and related to the ischial spine. ACOG has defined five stations above (-5) and below (+5) the level of the spine (0 stations). Minus five corresponds to the pelvic inlet, zero to the level of the ischial spine, and plus four corresponds to the pelvic floor.

Traditionally, labor progression has been assessed by digital examination of cervical dilatation and fetal descent. Recent studies, however, dispute these findings and found the clinical examination of fetal descent and position to be unprecise and subjective with a high interobserver variation. Dupuis et al. made an important contribution to this debate when he rigorously assessed the accuracy of station diagnosis with digital examinations. . This study provides evidence that digital assessment of fetal head station is unreliable.

However, a study from 2019 found a good correlation between clinical assessments and ultrasound examinations when only one experienced clinician and one trained ultrasound examiner compared their results.

In this study, we aim to evaluate the accuracy of and consistency between vaginal examination and transperineal ultrasound head station measurements.

ELIGIBILITY:
Inclusion Criteria:

* At or over 36 weeks pregnant women
* Pregnant women at the active phase of the first stage of labor
* Pregnant women at the second stage of labor

Exclusion Criteria:

* Breech presentation
* Fetal anomaly
* In utero ex fetus cases
* Trial of labor after cesarean cases
* Pregnant women at the latent phase of the first sage of labor

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Study Population: Pregnant women at 36 weeks or over gestational weeks at the active phase of the first stage and the second stage of labor.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-02-20 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Acuracy of the fetal head progression distance | At any time in active phase of first stage or second stage of labor
  Transperineal measurement of fetal head station will be compared with vaginal examination of fetal head descent and these two measurements correlated with delivery outcomes

SECONDARY OUTCOMES:
Interobserver agreement between vaginal examination fetal head station | At any time in active phase of first stage or second stage of labor
  The examination of fetal head levels by two clinicians compared with eachother.
Interobserver agreement between ultrasonographic fetal head station measurement | At any time in active phase of first stage or second stage of labor
  The correlation between two clinicians in measuring ultrasonographic fetal head station.

CONTACTS AND LOCATIONS:
Overall Officials: Murat Yassa, MD, Study Director — Specialist
Locations (1):
- Sehit Prof Dr Ilhan Varank Sancaktepe Training and Research Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Ciaciura-Jarno M, Cnota W, Wojtowicz D, Niesluchowska-Hoxha A, Ruci A, Kierach R, Stepien A, Nowak A, Sodowska P. Evaluation of selected ultrasonography parameters in the second stage of labor in prediction mode of delivery. Ginekol Pol. 2016;87(6):448-53. doi: 10.5603/GP.2016.0024. PMID 27418223
- [Background] Akmal S, Kametas N, Tsoi E, Hargreaves C, Nicolaides KH. Comparison of transvaginal digital examination with intrapartum sonography to determine fetal head position before instrumental delivery. Ultrasound Obstet Gynecol. 2003 May;21(5):437-40. doi: 10.1002/uog.103. PMID 12768552
- [Background] Ramphul M, Ooi PV, Burke G, Kennelly MM, Said SA, Montgomery AA, Murphy DJ. Instrumental delivery and ultrasound : a multicentre randomised controlled trial of ultrasound assessment of the fetal head position versus standard care as an approach to prevent morbidity at instrumental delivery. BJOG. 2014 Jul;121(8):1029-38. doi: 10.1111/1471-0528.12810. Epub 2014 Apr 11. PMID 24720273
- [Background] Dupuis O, Silveira R, Zentner A, Dittmar A, Gaucherand P, Cucherat M, Redarce T, Rudigoz RC. Birth simulator: reliability of transvaginal assessment of fetal head station as defined by the American College of Obstetricians and Gynecologists classification. Am J Obstet Gynecol. 2005 Mar;192(3):868-74. doi: 10.1016/j.ajog.2004.09.028. PMID 15746684
- [Background] Iversen JK, Jacobsen AF, Mikkelsen TF, Eggebo TM. Structured clinical examinations in labor: rekindling the craft of obstetrics. J Matern Fetal Neonatal Med. 2021 Jun;34(12):1963-1969. doi: 10.1080/14767058.2019.1651283. Epub 2019 Aug 19. PMID 31422727
- See also: World Health Organization. Intrapartum care for a positive childbirth experience. 2018. ISBN 978-92-4-155021-5 — https://apps.who.int/iris/bitstream/handle/10665/260178/9789241550215-eng.pdf
- See also: Brief History of Intrapartum Ultrasonography — https://link.springer.com/chapter/10.1007/978-3-030-57595-3_2